CLINICAL TRIAL: NCT06720051
Title: Efficacy of Intraosseous Versus Submucosal Dexamethasone Injection in Terms of Pain, Facial Swelling and Interincisal Opening Among Patients Undergoing Third Molar Surgery
Brief Title: Intraosseous Versus Submucosal Dexamethsone Injection in Third Molar Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Services Institute of Medical Sciences, Pakistan (Other Government)
Responsible Party: Principal Investigator, Mahreen Mahmood, OMFS Resident, Services Institute of Medical Sciences, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U1111-1315-4156
Record Dates: First submitted 2024-12-02; First posted 2024-12-06 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Third Molar Surgery
Keywords: intraosseous dexamethasone injection; submucosal dexamethasone injection; Third molar surgery; facial pain in third molar surgery; facial swelling in 3rd molar surgery; interincisal opening in third molar surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A will undergo intraosseous dexamethasone injection after 3rd molar surgery (Experimental): In Group A, patients will receive 4 mg dexamethasone intraosseous injection into the bone distal to the socket of impacted third molar immediately after extraction of the third molar and before suturing
  Interventions: Procedure: Intraosseous dexamethasone injection after 3rd molar surgery
- Group B will undergo submucosal dexamethasone injection after 3rd molar surgery (Active Comparator): In Group B, patients will receive 4 mg dexamethasone submucosal injection into the buccal vestibule opposite to the surgical site of impacted third molar immediately after surgery.
  Interventions: Procedure: Submucosal dexamethasone injection after 3rd molar surgery

INTERVENTIONS:
Procedure: Intraosseous dexamethasone injection after 3rd molar surgery — In Group A, patients will receive 4 mg dexamethasone intraosseous injection into the bone distal to the socket of impacted third molar immediately after extraction of the third molar and before suturing
  Arms: Group A will undergo intraosseous dexamethasone injection after 3rd molar surgery
Procedure: Submucosal dexamethasone injection after 3rd molar surgery — In Group B, patients will receive 4 mg dexamethasone submucosal injection into the buccal vestibule opposite to the surgical site of impacted third molar immediately after surgery.
  Arms: Group B will undergo submucosal dexamethasone injection after 3rd molar surgery

SUMMARY:
The goal of this clinical trial is to learn if intraosseous dexamethasone injection is better for pain and swelling postop 3rd molar surgery than submucosal dexamethasone injection. The main questions it aims to answer are:

Does intraosseous dexamethasone injection provide better pain relief and lessen facial swelling than submucosal dexamethasone injection Does intraosseous dexamethasone injection provide better interincisal opening than submucosal dexamethasone injection Researcher will compare both the techniques to see if intraosseous dexamethasone injection works better than submucosal dexamethasone injection

Participants will:

Be assessed at 3rd and 7th day postoperatively Pain will be assessed through visual analog scale score Facial measurement will be calculated as horizontal measurement plus vertical measurement divided by 2, where horizontal measurement will be taken as the distance between corner of the mouth and the earlobe attachment, and vertical measurement will be taken as distance from outer canthus of the eye to the angle of jaw.

Interincisal opening will be measured from the incisal edge of the maxillary central incisors to the incisal edge of mandibular central incisors at the midline by using millimeter ruler

DETAILED DESCRIPTION:
OBJECTIVE: To determine the efficacy of intraosseous versus submucosal dexamethasone injection in terms of pain, facial swelling and interincisal opening among patients undergoing mandibular 3rd molar surgery OPERATIONAL DEFINITIONS

Mandibular third molar:

A mandibular third molar prevented from erupting into position because of malposition or lack of space will be assessed on clinical (visual examination in oral cavity) and radiographical examination (periapical and/or orthopantomogram) by using Pell and Gregory classification method and modified Winter's classification method

Efficacy:

Efficacy of intraosseous and submucosal dexamethasone will be assessed in terms of lower VAS pain score, less facial swelling, and greater interincisal distance.

Pain:

Pain is an unpleasant sensory and emotional experience associated with, or resembling that associated with, actual or potential tissue damage. Pain will be assessed using visual analogue scale (VAS), which is a self-administered continuous scale comprised of a line of 10 cm in length, anchored by "no pain (score 0)" and "pain as bad as it could be (score 10)". The patient is asked to place a line perpendicular to the VAS line at the point that represents their pain intensity; and score is determined by measuring the distance between "no pain (score 0)" anchor and the patient's mark. A higher score indicates greater pain intensity

Interincisal opening:

Interincisal opening will be measured from the incisal edge of the maxillary central incisors to the incisal edge of mandibular central incisors at the midline by using millimeter ruler.

Facial swelling:

Facial swelling is the buildup of fluid in the tissues of the face. Facial measurement will be calculated as horizontal measurement plus vertical measurement divided by 2, where horizontal measurement will be taken as the distance between corner of the mouth and the earlobe attachment, and vertical measurement will be taken as distance from outer canthus of the eye to the angle of jaw.

These measurements will be taken as baseline measurement before the procedure, and then on day 3 and 7 after procedure.

HYPOTHESIS:

Intraosseous dexamethasone is more efficacious in terms of pain control, less facial swelling and greater interincisal opening than submucosal dexamethasone among patients undergoing mandibular third molar surgery.

MATERIAL AND METHODS

STUDY DESIGN:

Randomized controlled trial (RCT)

SETTINGS:

Department of Oral & Maxillofacial Surgery, Services Institute of Medical Sciences, Lahore

DURATION OF STUDY:

Six months after approval of synopsis

SAMPLE SIZE:

A sample size of 76 (38 in each group) calculated using the expected mean difference of pain VAS 0.9 between intraosseous dexamethasone group (3.3±1.3) and submucosal dexamethasone group (2.4±1.1) with 95.0% confidence level and 90.0% power of test.

Formula n = (Zα/2+Zβ)2 * _2 σ2_ d2 Where Zα/2 = Critical value of the normal distribution = 1.96 for 95.0% Cl Zβ = Critical value of the normal distribution = 1.28 for 90.0% power of test σ2 = Population variance = 1.44 d = Difference = 0.9

SAMPLING TECHNIQUE:

Non-probability consecutive sampling technique

DATA COLLECTION PROCEDURE:

The study will be approved by the Institutional Ethics Review Committee of Services Institute of Medical Sciences Lahore. All eligible patients undergoing mandibular third molar surgery will be invited to participate in the study and informed consent will be obtained from all volunteer participants. Total 76 patients (38 in each group) will be randomized into two equal-size groups i.e. Group A and Group B by lottery method. A structured proforma will be used to collect demographic and clinical data.

Before surgery, age, gender, Pell & Gregory type, Winter's type, baseline interincisal opening and facial measurement will be noted. In Group A, patients will receive 4 mg dexamethasone intraosseous injection into the bone distal to the socket of impacted third molar immediately after extraction of the third molar and before suturing. In Group B, patients will receive 4 mg dexamethasone submucosal injection into the buccal vestibule opposite to the surgical site of impacted third molar immediately after surgery. A team of supervisor and researcher will perform all these procedures. All patients will be prescribed tablet naproxium sodium 550mg twice a day for two days.

Patients will be assessed for pain, interincisal opening and facial measurement at day 3 and 7 after surgery. As per operational definitions, efficacy in terms of lower pain VAS score, less facial swelling, and greater interincisal opening will be compared between intraosseous and submucosal dexamethasone groups.

DATA ANALYSIS PROCEDURE:

Statistical Package for Social Sciences (SPSS) version 27 will be used for data entry and analysis. The quantitative variables such as age, interincisal opening, facial measurement and pain VAS score will be reported using mean ± standard deviation. The qualitative variables such as gender, Pell & Gregory type, and Winter's type will be reported using number (percent). The comparison between intraosseous and submucosal dexamethasone groups for interincisal opening, facial measurement and pain VAS score will be performed by t-test. The data will be stratified for age and gender. After stratification comparison between intraosseous and submucosal dexamethasone groups for interincisal opening, facial measurement and pain VAS score will be performed by t-test. P-value of ≤0.05 will be considered as significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing mandibular third molar surgery
* Age 18 to 35 years
* Male and female

Exclusion Criteria:

* Uncontrolled systemic medical problems including diabetes and hypertension
* Presence of any cyst, tumor, or other pathological condition in the molar area
* Presence of any craniofacial anomalies, congenital deformities or syndromes
* Patients with known adverse effects of steroid use
* Previous history of orthodontic treatment
* Have a pain disorder or taking pain medications
* Pregnant and lactating mothers

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Pain | 3rd and 7th day post operatively
  Pain is an unpleasant sensory and emotional experience associated with, or resembling that associated with, actual or potential tissue damage. Pain will be assessed using visual analogue scale (VAS), which is a self-administered continuous scale comprised of a line of 10 cm in length, anchored by "no pain (score 0)" and "pain as bad as it could be (score 10)". The patient is asked to place a line perpendicular to the VAS line at the point that represents their pain intensity; and score is determined by measuring the distance between "no pain (score 0)" anchor and the patient's mark. A higher score indicates greater pain intensity
Interincisal opening | 3rd and 7th day post operatively
  Interincisal opening will be measured from the incisal edge of the maxillary central incisors to the incisal edge of mandibular central incisors at the midline by using millimeter ruler
Facial swelling | 3rd and 7th day post operatively
  Facial swelling is the buildup of fluid in the tissues of the face. Facial measurement will be calculated as horizontal measurement plus vertical measurement divided by 2, where horizontal measurement will be taken as the distance between corner of the mouth and the earlobe attachment, and vertical measurement will be taken as distance from outer canthus of the eye to the angle of jaw

CONTACTS AND LOCATIONS:
Locations (1):
- Services Institute of Medical Sciences Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sirintawat N, Sawang K, Chaiyasamut T, Wongsirichat N. Pain measurement in oral and maxillofacial surgery. J Dent Anesth Pain Med. 2017 Dec;17(4):253-263. doi: 10.17245/jdapm.2017.17.4.253. Epub 2017 Dec 28. PMID 29349347